CLINICAL TRIAL: NCT03098940
Title: A Two Part, Open Label, Randomized, Four Period Cross-over Study to Compare the Bioavailability of Two Different Dronabinol Formulations in Healthy Male and Female Volunteers
Brief Title: A Bioavailability Study on Dronabinol
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Axim Biotechnologies (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MedChew
Record Dates: First submitted 2017-03-21; First posted 2017-04-04 (Actual); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: THC
MeSH Terms: interventions — Chewing Gum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Chewing gum (Experimental): Chewing gum with various doses of dronabinol
  Interventions: Drug: Chewing Gum
- Capsule (Marinol) (Active Comparator): Marinol is a product manufactured by AbbVie Capsule with various strengths of Marinol
  Interventions: Drug: Chewing Gum

INTERVENTIONS:
Drug: Chewing Gum — During the study healthy subjects will receive single doses of the various strengths of dronabinol

SUMMARY:
This study is a two part study

DETAILED DESCRIPTION:
This study is a two part, open label, randomized, four periods cross-over study with a washout of at least 1 week between subsequent dosing occasions

ELIGIBILITY:
Inclusion Criteria:

* Healthy, non-smoking male and female subject, aged between 18 and 55 year of age (inclusive) with a BMI ≥18.0 kg/m2 and ≤ 30.0 kg/m2.

Exclusion Criteria:

* Smokers

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-01 (Estimated); Primary Completion 2018-04 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Bioequivalence | up to 48 hours post-dose
  based on Peak Plasma Concentration (Cmax)
Bioequivalence | up to 48 hours post-dose
  based on Area under the plasma concentration versus time curve (AUC)

IPD SHARING:
Plan to Share IPD: No